CLINICAL TRIAL: NCT04292600
Title: Testing of Identification Markers for Stroke
Acronym: TIME
Status: Completed | Type: Observational
Sponsor: POCKiT diagnostics Ltd (Industry)
Collaborators: University of Alabama at Birmingham (Other); University of Mississippi Medical Center (Other); Bay Area Consulting Telemedicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: POCKiT
Record Dates: First submitted 2020-02-20; First posted 2020-03-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Stroke, Ischemic; Infarction, Middle Cerebral Artery; Infarction, Anterior Circulation, Brain
Keywords: large vessel occlusion strokes
MeSH Terms: conditions — Ischemic Stroke; Infarction, Middle Cerebral Artery; Brain Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BRH: Cohort recruited at Brandon Regional Hospital by Bay Area Consulting Telemedicine
  Interventions: Diagnostic Test: POCKiT diagnostics' algorithm for LVO detection

INTERVENTIONS:
Diagnostic Test: POCKiT diagnostics' algorithm for LVO detection — Measurement of blood biomarkers and integration within Pockit diagnostics' algorithm for LVO detection

SUMMARY:
Stroke is the third leading cause of death and the first cause of physical disability and dementia worldwide. Ischemic stroke caused by large vessel occlusion (LVO) is responsible for the vast majority of deaths and disabilities. A very effective and safe treatment, called mechanical thrombectomy (MT) is available for LVO patients. Nevertheless, no blood biomarkers able to identify LVO patients rapidly and to direct them to CT angiography and thrombectomy currently exist.

The TIME study is an observational prospective cohort study. All Patients referred to the emergency department or stroke unit with a suspected stroke as identified by paramedics, nurses or clinicians will be enrolled in the study. A panel of blood biomarkers will be analysed retrospectively via standard laboratory assays.

The main outcome of the TIME study will be the evaluation of the clinical diagnostic performance of a panel of blood biomarkers, in conjunction with clinical data, for the identification of large vessel occlusion ischemic stroke subtype. This study will allow the identification and evaluation of a final panel of biomarkers and will prompt the development of a test for LVO stroke diagnosis.

DETAILED DESCRIPTION:
Stroke affects 16M people in the world every year and 100K in the UK only. More than 30% of these patients die and 90% of survivors develop permanent disabilities as a consequence of stroke. There are two main types of stroke, ischemic and haemorrhagic. Ischemic stroke is caused by the formation of a clot in a blood vessel in the brain and represents ~85% of stroke patients. Haemorrhagic stroke is due to the rupture of a blood vessel in the brain, with consequent bleeding, and it represents ~15% of stroke patients. Both stroke subtypes cause brain damage and their symptoms are very similar. In addition to these two types of stroke, among the population of suspected stroke patients, there are the so-called stroke "mimics". These are conditions that appear with stroke-like symptoms (e.g. migraine, epilepsy, encephalitis, etc) but that are not stroke.

The deadliest stroke subtype is the one caused by occlusion of large vessels (LVO) in the brain. For these patients, a new treatment is available, called thrombectomy, which is a surgical procedure that mechanically removes the clot via a probe inserted at the level of the groin. Treatment of LVO patients with mechanical thrombectomy (MT) significantly increases the chances of survival, as well as decreases the extent of disability1. MT is only available in comprehensive stroke centres (CSC), and LVO patients have to be transported specifically to CSC in order to be treated and increase their chances of survival. MT has been proven a safe and effective treatment for LVO stroke until 24 hours from stroke onset2, indicating that detection of LVO strokes several hours after onset can significantly aid the stroke care pathway.

Current treatment of stroke patients is dependent on diagnosis via computerised tomography (CT) scan to the head. CT is highly accurate for detection of brain haemorrhages, but is very inaccurate for detection of ischemic stroke or LVOs3. In case of a negative result from CT, neurologists can order a further MRI scan to confirm ischemic stroke. If LVO is suspected, patients are transported to the nearest CSC where a further procedure, called CT angiography, is performed. The identification of LVO patients can be a very lengthy process that wastes precious time and makes stroke patients worse.

Fast diagnosis of stroke patients at their first point of admission (i.e. ambulance or emergency department) able to identify LVO patients could quickly direct patients to CSC and significantly improve treatment of the most dangerous stroke subtype. Several studies have investigated the ability of pre-hospital assessment scores based on patient symptoms to be performed in the ambulance4-7. Despite this, these scoring scales lack the accuracy required for triaging LVO patients with confidence. A more accurate diagnostic test able to complement these assessment scores and direct LVO patients to CSC and CT angiography is much needed8.

POCKiT DX are developing a novel device for stroke diagnosis that combines accurate blood biomarkers with ultra-rapid (<20 minutes) biomarker detection within a point-of-care device. The panel of blood biomarkers identified by POCKiT DX was tested in 80 patients with suspected stroke and accuracy of 83% (CI 95%: 74-92%), sensitivity of 86% (CI 95%: 74-98%), and specificity of 82% (CI 95%: 68-95%) was observed for LVO identification.

The aim of the TIME study is to evaluate the clinical diagnostic performance of a panel of blood biomarkers identified by POCKiT diagnostics in the identification of LVO stroke patients among the population of suspected stroke. Diagnostic performance of blood biomarkers alone, and in conjunction with clinical data, including pre-hospital stroke assessment scores (e.g. EMSA), will be evaluated. Results of this study will direct the development of a diagnostic test for directing stroke patients to the right treatment, more rapidly, improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the ambulance or emergency department for suspected stroke.
* Time from stroke onset < 18 hours

Exclusion Criteria:

* Received thrombolytic therapy (e.g. tPA, Alteplase) before collection of blood;
* (Anticipated) inability to provide a blood sample;
* Time from stroke onset > 18 hours.
* At time of consent participating in a Clinical Trial Investigational Medicinal Product (CTIMP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ambulance and ED with suspected stroke will be recruited in the study. Patient population is expected to be composed of ~50% ischemic strokes (of which ~30-40% could have LVOs), ~40% stroke mimics, and ~10% haemorrhagic strokes.
Sampling Method: Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy measures for LVO detection vs non-LVO stroke activations | 1 year
  Accuracy of pre-defined algorithm thresholds for LVO identification from the population of all suspected strokes (Ischemics non-LVO, Hemorrhagic, Mimics, TIAs)

SECONDARY OUTCOMES:
Optimisation of the cut-off points of the diagnostic algorithm for LVO detection | 1 year
  Determine optimal cut-off points for diagnostic algorithm for detection of LVO vs non-LVO

CONTACTS AND LOCATIONS:
Overall Officials: Shashank Shekar, MD, Principal Investigator — University of Mississippi Medical Center; Toby Gropen, MD, Principal Investigator — University of Alabama in Birmingham Comprehensive Stroke Center; Allauddin Khan, MD, Principal Investigator — BAC Telemed (Brandon Regional Hospital)
Locations (3):
- United States (3):
  - University of Alabama in Birmingham Comprehensive Stroke Center, Birmingham, Alabama
  - BAC Telemed - Brandon Regional Hospital, Brandon, Florida
  - University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malhotra K, Gornbein J, Saver JL. Ischemic Strokes Due to Large-Vessel Occlusions Contribute Disproportionately to Stroke-Related Dependence and Death: A Review. Front Neurol. 2017 Nov 30;8:651. doi: 10.3389/fneur.2017.00651. eCollection 2017. PMID 29250029
- [Background] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157
- [Background] Gropen TI, Boehme A, Martin-Schild S, Albright K, Samai A, Pishanidar S, Janjua N, Brandler ES, Levine SR. Derivation and Validation of the Emergency Medical Stroke Assessment and Comparison of Large Vessel Occlusion Scales. J Stroke Cerebrovasc Dis. 2018 Mar;27(3):806-815. doi: 10.1016/j.jstrokecerebrovasdis.2017.10.018. Epub 2017 Nov 22. PMID 29174289
- [Derived] Durrani Y, Gerstl JVE, Murphy D, Harris A, Saali I, Gropen T, Shekhar S, Kappel AD, Patel NJ, Du R, Guardia REA, Vicenty-Padilla JC, Dmytriw AA, Pereira VM, Izzy S, Khan A, Aziz-Sultan MA, Liebeskind DS, Davies JM, Siddiqui AH, Gaude E, Bernstock JD. Prospective Validation of Glial Fibrillary Acidic Protein, d-Dimer, and Clinical Scales for Acute Large-Vessel Occlusion Ischemic Stroke Detection. Stroke Vasc Interv Neurol. 2024 May 17;4(4):e001304. doi: 10.1161/SVIN.123.001304. eCollection 2024 Jul. PMID 41585381

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT04292600/Prot_SAP_002.pdf
  • Informed Consent Form (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT04292600/ICF_000.pdf